CLINICAL TRIAL: NCT07017868
Title: Correlation Between Serum Uric Acid, Serum Homocysteine Level and Interleukin- 17 in Lupus Nephritis Patients
Status: Recruiting | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Sara Mohamed Ahmed, resident-clinical pathology sohag university hospital, Sohag University
Other Study IDs: Soh-Med--25-4-07MS
Record Dates: First submitted 2025-06-04; First posted 2025-06-12 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Homocysteine Level and Interleukin- 17 in Lupus Nephritis Patients

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- CASE 1: Patient with systemic lupus witout nephritis
  Interventions: Diagnostic Test: interleukin- 17
- case 2: Patient with systemic lupus with nephritis
  Interventions: Diagnostic Test: interleukin- 17
- controls: healthy people
  Interventions: Diagnostic Test: interleukin- 17

INTERVENTIONS:
Diagnostic Test: interleukin- 17 — focused on the importance of IL-17 in SLE, and its relation to different disease activity

SUMMARY:
Systemic lupus erythematosus (SLE) is a chronic inflammatory multisystem autoimmune disease characterized by pathogenic autoantibodies production against nuclear structures . SLE affecting mainly women of childbearing age and is characterized by unpredictable flares and remissions. Disease severity varied from a mild episodic disorder to a rapidly progressive life-threatening illness. The kidney is the most commonly involved visceral organ in SLE. Therefore, identifying new noninvasive biomarkers of LN severity and outcome is mandatory. IL-17 is a potent pro-infammatory cytokine that amplifes T-cell activation and stimulates fibroblast cells, endothelial, and epithelial cells to produce several pro-infammatory mediators, including IL-1β, IL-6, and TNF-α. IL-17 receptor signaling enhances the expression of multiple pro-infammatory mediators. Hence, IL-17 enhances the production of neutrophil-attracting chemokines

DETAILED DESCRIPTION:
Systemic lupus erythematosus (SLE) is a chronic inflammatory multisystem autoimmune disease characterized by pathogenic autoantibodies production against nuclear structures. SLE affecting mainly women of childbearing age and is characterized by unpredictable flares and remissions. Disease severity varied from a mild episodic disorder to a rapidly progressive life-threatening illness. The kidney is the most commonly involved visceral organ in SLE Lupus nephritis (LN) is one of the most serious manifestations of SLE since it is associated with significant morbidity and mortality and affects up to 60% of SLE patients. Nephritic syndrome and acute kidney injuries can complicate LN and increase the risk of end stage renal disease (ESRD) . Early diagnosis of renal involvement in SLE patients is important to improve the long-term outcome and increase the survival rate .

LN is diagnosed by either the presence of proteinuria (>0.5 g/day), active urinary sediment (with red blood cell, granular, tubular and/or mixed casts), or an unexplained rise in serum creatinine. A renal biopsy is known to be the gold standard for the diagnosis of LN because it gives information and details about the pattern and severity of kidney affection as well as the exclusion of other mimics of LN . Each of these factors weighs heavily on treatment choices. However, kidney biopsy is an invasive technique, and it is contraindicated in some situations such as bleeding and infection, associated with renal biopsy .

Therefore, identifying new noninvasive biomarkers of LN severity and outcome is mandatory. IL-17 is a potent pro-infammatory cytokine that amplifes T-cell activation and stimulates fibroblast cells, endothelial, and epithelial cells to produce several pro-infammatory mediators, including IL-1β, IL-6, and TNF-α. IL-17 receptor signaling enhances the expression of multiple pro-infammatory mediators. Hence, IL-17 enhances the production of neutrophil-attracting chemokines .

Few studies focused on the importance of IL-17 in SLE, particularly LN, and its relation to different disease activity parameters, so we aimed to explore its relation with uric acid and homocysteine in LN.

Also, Lupus nephritis (LN) is closely associated with hyperuricemia, and uric acid is the metabolite of purine that is excreted mainly in urine and considered a risk factor for renal involvement in systemic lupus erythematosus (SLE).

We postulated that patients with lupus nephritis are more likely to have elevated homocysteine levels. Homocysteine is metabolized by two alternative pathways, including its remethylation and transsulfuration. Elevated serum homocysteine can occur in 5 to 10 percent of the population. Increased serum homocysteine levels are seen in approximately 15% of patients with systemic lupus erythematosus.

ELIGIBILITY:
Inclusion Criteria:

* ● Aged ≥18 years.

  * SLE patients fulfilling the SLE International Collaborating Clinics (SLICC) classification criteria and matched controls.
  * Patients cooperative and can answer questions.
  * Patients who are able and willing to give written informed consent

Exclusion Criteria:

* ● Individuals with other autoimmune diseases.

  * Patients receive any hyperuricemia treatment
  * Pregnancy
  * Malignancy
  * Diabetes.
  * Hypertension.
  * Heart failure.
  * Hepatic diseases.
  * Chronic renal failure other than lupus nephritis.
  * Renal artery stenosis.
  * Renal vein thrombosis.
  * Intrarenal arteriovenous fistula.
  * Obstructive nephropathy.
  * Urinary tract obstruction that could affect RI of intra renal arteries.
  * Uncooperative patients.
  * Patients not able and willing to give written informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This study will include 80 established SLE patients who will be recruited from Rheumatology and Rehabilitation department at Sohag university hospital,40 of them with nephritis and other 40 witout nephritis, in addition to 40 control who will be matched for sex, age, and level of schooling without history of any systemic active disease (healthy people).
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
SLE disease activity index (SLEDAI) will be assessed | 1 year
  . IL-17 is a potent pro-infammatory cytokine that amplifes T-cell activation and stimulates fibroblast cells, endothelial, and epithelial cells to produce several pro-infammatory mediators, including IL-1β, IL-6, and TNF-α. IL-17 receptor signaling enhances the expression of multiple pro-infammatory mediators

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag university Hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Alforaih N, Whittall-Garcia L, Touma Z. A Review of Lupus Nephritis. J Appl Lab Med. 2022 Oct 29;7(6):1450-1467. doi: 10.1093/jalm/jfac036. PMID 35932197
- [Background] Zhu S, Qian Y. IL-17/IL-17 receptor system in autoimmune disease: mechanisms and therapeutic potential. Clin Sci (Lond). 2012 Jun;122(11):487-511. doi: 10.1042/CS20110496. PMID 22324470
- [Background] Ameer MA, Chaudhry H, Mushtaq J, Khan OS, Babar M, Hashim T, Zeb S, Tariq MA, Patlolla SR, Ali J, Hashim SN, Hashim S. An Overview of Systemic Lupus Erythematosus (SLE) Pathogenesis, Classification, and Management. Cureus. 2022 Oct 15;14(10):e30330. doi: 10.7759/cureus.30330. eCollection 2022 Oct. PMID 36407159
- [Background] Anstee QM, Castera L, Loomba R. Impact of non-invasive biomarkers on hepatology practice: Past, present and future. J Hepatol. 2022 Jun;76(6):1362-1378. doi: 10.1016/j.jhep.2022.03.026. PMID 35589256